CLINICAL TRIAL: NCT06904846
Title: Prospective Post-market Clinical Follow-up (PMCF) Study Aimed to Evaluate the Change in Glucometric Parameters in Adult Patients With Type 1 or Type 2 DiabETes From Europe Using the iCan o3 CGM SysTem for a 60-day Period
Brief Title: To Evaluate the Change in Glucose Parameters in Adult Patients With Type 1 or Type 2 Diabetes From Europe Using the iCan o3 CGM System for 60 Days Period
Acronym: DETECT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sinocare (Industry)
Collaborators: Archer Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPI031-PMCFR-001
Record Dates: First submitted 2025-03-17; First posted 2025-04-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus; Continuous Glucose Monitoring System
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Type 1 diabetes (T1D) or Type 2 diabetes (T2D) (Experimental): The start-up pathway is for all persons with T2D who are not being treated in another diabetes system. People with T2D in remission can also apply for the start-up pathway. The care pathway is for persons with T2D who are treated with Glucagon-like peptide-1 (GLP-1) analogues (injectable or pill) or 1 to 2 insulin injections/day. This pathway can also be initiated if treatment with blood sugar-lowering medication (pills) is insufficient and a GLP-1 analogue or insulin is being considered. The diabetes convention is intended for those in need of specialist management (T1D patients and a limited group of T2D patients on intensive insulin therapy (3 to 4 times a day)), given complex insulin therapy.
  Interventions: Device: iCan o3 CGM Continuous Glucose Monitoring System

INTERVENTIONS:
Device: iCan o3 CGM Continuous Glucose Monitoring System — A continuous Glucose Monitoring System (CGM System) is a real-time, continuous glucose monitoring device indicated for the management of diabetes for adult persons (age 18 and older). It is intended to replace finger prick blood glucose testing for diabetes treatment decisions. The CGM System also shows trends and tracks patterns, and aids in the detection of episodes of hyperglycemia and hypoglycemia, facilitating both acute and long-term therapy adjustments. Interpretation of the CGM System results should be based on the glucose trends and several sequential readings over time.
  The CGM System can be used in conjunction with smart devices with corresponding applications (apps) where the user manually controls actions for therapy decisions. During this study, Self-Monitoring Blood Glucose (SMBG) assessed by an iCan o3 CGM System blinded to the patient for 15 days as the baseline and unblinded observation period using an iCan o3 CGM System for 45 days occurs.

SUMMARY:
This study is a post-market, prospective, interventional, multicenter clinical trial designed to evaluate the impact of the iCan O3 Continuous Glucose Monitoring (CGM) System on glycemic control in adults with Type 1 (T1D) or Type 2 Diabetes (T2D). Coordinated by Prof. Dr. Christophe De Block at Universitair Ziekenhuis Antwerpen (UZA), Belgium, and sponsored by Changsha Sinocare Inc., the study aims to assess changes in glucometric parameters over 60 days. The primary objective is to demonstrate an improvement in Time in Range (TIR) compared to baseline, measured during an initial 15-day blinded period using self-monitored blood glucose (SMBG) assessed by the iCan O3 CGM System. Secondary objectives include evaluating the system's efficacy, safety, and usability and patient-reported outcomes such as treatment satisfaction and diabetes management impact. The study will enroll 70 patients aged 18-75 with HbA1c >7.5%, stable treatment regimens, and smartphone proficiency while excluding individuals with recent diabetes-related hospitalizations, severe comorbidities, or conflicting trial participation. The study timeline spans from February 2025 to September 2025, with patients undergoing a 15-day blinded period followed by a 45-day unblinded period where real-time CGM data is accessible. Key endpoints include improvements in TIR, Time Below Range (TBR), Time Above Range (TAR), mean glucose levels, glucose variability, and patient-reported outcomes and safety metrics such as device deficiencies and adverse events. Risks, including skin irritation and delayed glucose readings, will be mitigated through patient training and safety protocols. Anticipated benefits include improved glycemic control, reduced reliance on fingerstick testing, and enhanced quality of life. Data will be collected from CGM metrics, questionnaires, and adverse event logs, with statistical analysis comparing baseline and post-intervention outcomes. The study adheres to ethical standards and EU MDR 2017/745 regulations, aiming to validate the iCan O3 CGM System's clinical utility in real-world diabetes management.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age is between 18 and 75 years old. Patient age is between 18 and 75 years old.
2. Patient is clinically diagnosed with diabetes for at least 6 months (all treatment modalities are allowed).
3. Patient has a Hemoglobin A1c (HbA1c) of > 7,5%.
4. Patient is sensor naive.
5. Patient is willing to wear the device on the abdomen for the whole study period.
6. Patient has a stable (unchanged) treatment regimen for at least 3 months. "Stable treatment regimen" is considered no changes in prescribed number of insulin deliveries a day, and a change in total daily insulin dose of less than 10%. Patients currently taking glucagon-like peptide-1 (GLP1) analogs before the study can be included.
7. Patient has a compatible smartphone.
8. Patient shows sufficient skills using a smartphone and apps, as judged by the investigator.
9. Patient and investigator signed and dated the informed consent form prior to first sensor placement.

Exclusion Criteria:

1. Patient was hospitalized because of hyperglycemia/ketoacidosis within the last 6 months.
2. Patient was hospitalized because of hypoglycemia within the last 6 months.
3. Patient has a condition which may predispose him/her to hypoglycemia including, but not limited to, thyroid disease which is not well controlled, adrenal insufficiency, high dose steroid use in recent past or planned during study, significant renal or liver disease.
4. Patient has a planned magnetic resonance imaging (MRI), Computed Tomography (CT) scan or diathermic procedure during the period of sensor wear.
5. Patient with a significant medical or psychiatric disorder, or use of a medication which will affect the application of the protocol judged by the investigator.
6. Patient with cognitive difficulties that may impair the ability to follow the protocol judged by the investigator.
7. Patient is critically ill.
8. Patient has a coagulation disorder or takes heparin-like antiplatelet medication.
9. Patient is pregnant or is intending to become pregnant during the study period.
10. Patient does not take clinically acceptable contraception or does not practice abstinence.
11. Patient has a history of skin adhesive tolerance issues in the area of sensor placement.
12. Patient has abnormal skin at the anticipated glucose sensor insertion sites (excessive hair, burn, inflammation, infection, rash, and/or tattoo).
13. Patient has any medical history of malignant melanoma or breast cancer.
14. Patient has a medical history of any other cancers within the last five years except adequately treated basal cell or squamous carcinoma of the skin, or cervical carcinoma in-situ.
15. Patient has a history of alcohol or drug abuse within the last year.
16. Patient has a history of a seizure disorder.
17. Patient has a medical history of stroke, transitory cerebral ischemia, myocardial infarction, unstable angina or heart failure with in the past 12 months.
18. Patient is on dialysis.
19. Patient is implanted with a pacemaker.
20. Patient is currently being treated with drugs known to have significant interference with glucose metabolism, such as systemic corticosteroids, as judged by the investigator.
21. Patient has a concomitant pathology that might cause edema at the insertion sites (such as heart failure, liver failure, kidney failure defined as estimated Glomerular Filtration Rate (eGFR) <30 mL/min [stage ≥4]).
22. Patient underwent beta-cell transplantation.
23. Patient is unable / unwilling to provide informed consent.
24. Patient is unable to comply with the protocol or proposed study visits.
25. Patient who is currently enrolled in another clinical study, or has recently participated in a clinical study, that could potentially interfere with the outcomes or introduce bias into the results of the current study (as determined by the investigator). This includes studies involving investigational drugs, medical devices, or other interventions that could impact the safety, efficacy, or scientific integrity of this study.
26. Other reasons that require the investigator to exclude the patient from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of Glycemic control | 60 days
  The increased percentage of Time in range (TIR) compare to the baseline period

CONTACTS AND LOCATIONS:
Locations (1):
- UZA ANTWERP UZA Dienst Endocrinologie, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No